CLINICAL TRIAL: NCT06757387
Title: A Phase I/II, Open-Label, Single-Arm Study of Chidamide in Combination With Golidocitinib in Patients With Relapsed or Refractory Peripheral T-Cell Lymphoma
Brief Title: Chidamide Plus Golidocitinib in Relapsed/Refractory Peripheral T-Cell Lymphoma
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Peking University Cancer Hospital & Institute (Other)
Responsible Party: Principal Investigator, Yuqin Song, MD, Yuqin Song, MD, Director of Hematology Department, Peking University Cancer Hospital & Institute
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CSIIT-T42
Record Dates: First submitted 2024-12-13; First posted 2025-01-03 (Actual); Last update posted 2025-01-03 (Actual); Status verified 2025-01

CONDITIONS: Peripheral T-cell Lymphoma
Keywords: PTCL
MeSH Terms: conditions — Lymphoma, T-Cell, Peripheral | interventions — N-(2-amino-5-fluorobenzyl)-4-(N-(pyridine-3-acrylyl)aminomethyl)benzamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Combination Treatment Group (Experimental): Dose Level 1 (chidamide 20 mg BIW / golidocitinib 150 mg QD), Dose Level 0 (chidamide 20 mg BIW / golidocitinib 150 mg QOD) will be further investigated. If the MTD is not established after escalating to Dose Level 2 (chidamide 25 mg BIW / golidocitinib 150 mg QD)
  Interventions: Drug: chidamide and golidocitinib

INTERVENTIONS:
Drug: chidamide and golidocitinib — Enrolled patients will receive combination therapy with golidocitinib (150 mg QD or 150 mg QOD) and chidamide (20 mg BIW or 25 mg BIW)； If the MTD is determined at Dose Level 1 (chidamide 20 mg BIW / golidocitinib 150 mg QD), Dose Level 0 (chidamide 20 mg BIW / golidocitinib 150 mg QOD) will be further investigated. If the MTD is not established after escalating to Dose Level 2 (chidamide 25 mg BIW / golidocitinib 150 mg QD), the recommended Phase 2 dose (RP2D) will be determined through investigator consensus.

SUMMARY:
This is a Phase I/II, open-label, single-arm study investigating the combination of chidamide and golidocitinib in patients with relapsed or refractory peripheral T-cell lymphoma (PTCL). The Phase I portion utilizes a 3+3 dose-escalation design to determine the maximum tolerated dose (MTD) and recommended Phase 2 dose (RP2D) of the drug combination. The Phase II portion will then evaluate the efficacy and safety of the RP2D in approximately 28 patients with relapsed or refractory PTCL. Treatment will continue until disease progression, unacceptable toxicity, withdrawal of consent, or meeting other stopping criteria. The primary goal of Phase I is to establish the safety and MTD and the RP2D. The primary goal of Phase II is to evaluate the treatment efficacy and safety of the combination at RP2D.

DETAILED DESCRIPTION:
Phase I Study:

The Phase I study will enroll an estimated 6 to 12 subjects. Using a 3+3 dose-escalation design, three dose levels of chidamide and golidocitinib will be explored. Enrolled patients will receive combination therapy with golidocitinib (150 mg QD or 150 mg QOD) and chidamide (20 mg BIW or 25 mg BIW), according to enrollment time. Starting with the lowest dose level, three patients will be treated at each dose level and observed for toxicity during the first cycle. If no dose-limiting toxicity (DLT) is observed, the next higher dose level will be investigated. If one DLT is observed, an additional three patients will be treated at that dose level. Dose escalation will continue if no further DLTs are observed in these additional patients, but will terminate if a DLT occurs. If more than one DLT occurs among the initial three patients, dose escalation will terminate. The dose level immediately below that at which the DLT is determined will be established as the maximum tolerated dose (MTD).

If the MTD is determined at Dose Level 1 (chidamide 20 mg BIW / golidocitinib 150 mg QD), Dose Level 0 (chidamide 20 mg BIW / golidocitinib 150 mg QOD) will be further investigated. If the MTD is not established after escalating to Dose Level 2 (chidamide 25 mg BIW / golidocitinib 150 mg QD), the recommended Phase 2 dose (RP2D) will be determined through investigator consensus. Each subject will receive only one dose level and schedule during the study. After completion of the treatment period, subjects will enter the follow-up period.

Phase II Study:

The Phase II study is expected to enroll approximately 28 patients with relapsed or refractory peripheral T-cell lymphoma (PTCL). Patients will receive treatment with golidocitinib and chidamide. The doses of chidamide and golidocitinib will be the RP2D established in the Phase I study. Each treatment cycle will be 21 days in duration. Subjects will continue to receive treatment per the investigator's assessment, until documented disease progression, intolerable toxicity, withdrawal of consent, or if the subject meets other criteria for treatment discontinuation (whichever occurs first).

ELIGIBILITY:
Inclusion Criteria:

* The subject must fully understand the study, voluntarily participate, and sign an informed consent form.
* The subject must be ≥ 18 years of age and ≤ 80 years of age, of either sex.
* The subject must have a histopathologically confirmed diagnosis of peripheral T-cell lymphoma (PTCL) according to the 2016 WHO classification, including peripheral T-cell lymphoma not otherwise specified (PTCL-NOS), angioimmunoblastic T-cell lymphoma (AITL), NK/T-cell lymphoma, anaplastic large cell lymphoma ALK-positive (ALCL ALK+), anaplastic large cell lymphoma ALK-negative (ALCL ALK-), enteropathy-associated T-cell lymphoma, and hepatosplenic T-cell lymphoma.
* The subject must have relapsed or refractory disease following prior systemic therapy (including autologous hematopoietic stem cell transplantation). Note: The subject must have received ≥1 and ≤3 prior lines of systemic therapy. Relapsed is defined as recurrence following a CR. Refractory is defined as disease with stable disease (SD) or progressive disease (PD) during interim efficacy assessment with prior systemic chemotherapy, or failure to achieve a CR at the end of treatment and need for further therapy.
* The subject must have at least one evaluable or measurable lesion according to the Lugano 2014 criteria:Lymph node lesions: Measurable lymph nodes must have a long axis >1.5 cm.

Non-lymph node lesions: Measurable extranodal lesions must have a long axis >1.0 cm.

* The subject must have an Eastern Cooperative Oncology Group (ECOG) performance status of 0-2.
* The subject must meet the following laboratory criteria:

Absolute neutrophil count (ANC) ≥ 1.5 × 10^9/L. Platelet count (PLT) ≥ 100 × 10^9/L (≥ 50 × 10^9/L if with bone marrow infiltration).

Hemoglobin (HB) ≥ 80 g/L. Serum total bilirubin (TBIL) ≤ 1.5 times the upper limit of normal (ULN). Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 2.5 times the ULN.

Serum creatinine (Scr) ≤ 1.5 times the ULN.

* The subject must not have received any radiotherapy, chemotherapy, targeted therapy, or hematopoietic stem cell transplantation within 3 weeks prior to enrollment.
* The investigator must determine that the subject has a life expectancy of at least 6 months.

Exclusion Criteria:

* Subjects with central nervous system (CNS) involvement and/or concomitant hemophagocytic lymphohistiocytosis (HLH).
* Prior treatment with a JAK inhibitor (e.g., golidocitinib).
* Prior treatment with an HDAC inhibitor within 3 weeks before the start of study treatment.
* Impaired cardiac function or significant cardiac disease, including, but not limited to:

Myocardial infarction, congestive heart failure, or viral myocarditis within 6 months prior to screening; symptomatic cardiac disease requiring medical intervention, such as unstable angina or arrhythmia.

Cardiac functional class ≥ III (New York Heart Association (NYHA) functional classification).

Ejection fraction (EF) less than 50% or below the lower limit of normal of the study site's standard by echocardiogram.

A history of persistent cardiomyopathy. QT corrected by Fridericia's formula (QTcF) > 450 milliseconds, or a congenital long QT syndrome.

* Hepatitis B (positive hepatitis B surface antigen or positive hepatitis B core antibody) or Hepatitis C (positive HCV antibody or HCV-RNA titer above the upper limit of normal at the study site).
* Uncontrolled active infection (viral, bacterial, fungal, etc., such as infectious pneumonia) or a requirement for non-oral anti-infective treatment.
* Major surgery within 4-6 weeks prior to screening or scheduled major surgery during the study.
* Uncontrolled hypertension at screening, uncontrolled diabetes at screening.
* A history of active visceral bleeding within 3 months prior to screening.
* History of malignancy within the past 5 years that may interfere with protocol implementation or results analysis (with the exception of treated basal cell skin cancer, cervical carcinoma in situ, breast carcinoma in situ, in situ gastrointestinal mucosal cancer, and localized prostate cancer).
* a) Post solid organ transplant. b). A history of allogeneic hematopoietic stem cell transplantation.
* History of psychiatric illness or cognitive impairment.
* A history of drug abuse (non-medical use of narcotic drugs or psychotropic drugs) and a history of drug dependence (sedatives, hypnotics, analgesics, narcotics, stimulants, and psychomimetic drugs, etc.).
* Women who are pregnant or breastfeeding, or women of childbearing potential (WOCBP) or male patients whose partners are unwilling or unable to use effective methods of contraception for the duration of the study and for 12 weeks after the last dose of the study drug. [WOCBP includes: any woman who has experienced menarche and has not undergone successful surgical sterilization (hysterectomy, bilateral tubal ligation, or bilateral oophorectomy) or is not postmenopausal.
* Any condition that, in the opinion of the investigator, would make the subject unsuitable for the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2024-12-30 (Estimated); Primary Completion 2028-12-30 (Estimated); Study Completion 2030-12-30 (Estimated)

PRIMARY OUTCOMES:
dose-limiting toxicities (DLTs) | within 28 days
  A Dose-Limiting Toxicity (DLT) is defined as any of the following events that occur within the first cycle of combination therapy and are considered possibly related (including definitely related, probably related) to the investigational drug(s):
  Grade 4 neutropenia lasting for more than 5 days. Grade ≥3 neutropenia with fever (neutrophil count <1.0 × 10^9/L with a single temperature >38.3°C or a temperature ≥38°C lasting for more than 1 hour).
  Grade 4 thrombocytopenia or Grade 3 thrombocytopenia with a bleeding tendency. Grade 4 anemia. Grade 3 nausea or vomiting persisting for more than 48 hours despite antiemetic treatment.
  Grade 4 nausea or vomiting. Grade ≥3 QTc prolongation or Grade ≥2 other cardiac toxicity. Grade ≥3 non-hematologic toxicity (excluding nausea and vomiting that is not responsive to treatment).
  Treatment delay of more than 2 weeks in cycle 2 due to tolerability issues. Other: Clinically significant, intolerable toxicities, determined by investigator discussion t

SECONDARY OUTCOMES:
objective response rate (ORR) | within 12 months
  Objective response rate (ORR) based on CT images,ORR is calculated by adding the number of patients who achieve a Complete Response (CR) to the number of patients who achieve a Partial Response (PR).

IPD SHARING:
Plan to Share IPD: No